CLINICAL TRIAL: NCT02232035
Title: Intravenous Injection of Diazepam at the Beginning of Active Phase of Labor
Brief Title: Diazepam at the Active Phase of Labor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yunhai Chuai, Department of Obstetrics and Gynecology, Navy General Hospital, Beijing, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: chuaiyunhai-002
Record Dates: First submitted 2014-08-30; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Pain; Prolonged Labour
Keywords: diazepam; active phase
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal saline, active phase of labor (Placebo Comparator): A single dose intravenous injection of normal saline (2ml) at the beginning of active phase of labor in the group.
  Interventions: Drug: normal saline/diazepam at the active phase of labor
- diazepam, active phase of labor (Experimental): A single dose intravenous injection of diazepam (10mg, 2ml) at the beginning of active phase of labor in the group.
  Interventions: Drug: normal saline/diazepam at the active phase of labor

INTERVENTIONS:
Drug: normal saline/diazepam at the active phase of labor — A single dose intravenous injection of normal saline (2ml)/diazepam (10mg, 2ml) at the beginning of active phase of labor.

SUMMARY:
Prolonged labour can lead to increased maternal and neonatal mortality and morbidity due to increased risks of maternal exhaustion, postpartum haemorrhage and sepsis, fetal distress and asphyxia and requires early detection and appropriate clinical response. The risks for complications of prolonged labour are much greater in poor resource settings. Active management of labour versus physiological, expectant management, has shown to decrease the occurrence of prolonged labour. Administering sedatives during labour could also lead to faster and more effective dilatation of the cervix. Interventions to shorten labour, such as sedatives, can be used as a preventative or a treatment strategy in order to decrease the incidence of prolonged labour. As the evidence to support this is still largely anecdotal around the world. (Cochrane Database of Systematic Reviews 2013,CD009243.pub3.; Cochrane Database of Systematic Reviews 2012, CD009223.pub2.)

Hypothesis: Diazepam reduced the duration of labor and the severity of pain in labor.

ELIGIBILITY:
Inclusion Criteria:

* primigravida
* at term
* singleton pregnancy
* cephalic presentation
* spontaneous labour
* intact membranes at the beginning of active phase

Exclusion Criteria:

* induced labour
* spontaneous rupture of membranes at randomisation
* obstetric complications, or medical complications
* previous uterine scarring, or cervical surgery
* cervical dilatation of more than 5 cm
* other antispasmodics in the first stage
* malpresentation, macrosomia, cephalopelvic disproportion

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Duration of labor | labor
  Duration of first stage of labor. Duration of second stage of labour. Duration of third stage of labor. Total duration of labor.

SECONDARY OUTCOMES:
Rate of cervical dilatation | at the active phase of labor
Pain relief | every 30 minutes during the 3-hour period after administration of the trial drug
  Pain severity during the last contraction was assessed using a Visual Analogue Scale (VAS) (with anchor points of 0 = no pain at all and 10 = the most excruciating pain) every 30 minutes during the 3-hour period after administration of the trial drug. This information was used to derive measures of pain relief at each time-point using absolute change in pain intensity (on a 10-cm VAS) from pre-analgesia (baseline). In addition to analysing all the time-points together (as described in the section on statistical analysis), a specific analysis of pain relief at 60 minutes was conducted, because it was anticipated that the maximum analgesic effect would occur then. (Wee MYK, Tuckey JP, Thomas PW, Burnard S. A comparison of intramuscular diamorphine and intramuscular pethidine for labour analgesia: a two-centre randomised blinded controlled trial. BJOG 2014;121:447-456.)
Type of delivery | post partum, immediately

OTHER OUTCOMES:
Maternal adverse events | two weeks after childbirth
Neonatal adverse events | two weeks after childbirth
Maternal satisfaction | post partum, immediately

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Wang, Dr, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Rohwer AC, Khondowe O, Young T. Antispasmodics for labour. Cochrane Database Syst Rev. 2013 Jun 5;2013(6):CD009243. doi: 10.1002/14651858.CD009243.pub3. PMID 23737030
- [Result] Othman M, Jones L, Neilson JP. Non-opioid drugs for pain management in labour. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD009223. doi: 10.1002/14651858.CD009223.pub2. PMID 22786524
- [Result] Davies JM, Rosen M. Intramuscular diazepam in labour. A double-blind trial in multiparae. Br J Anaesth. 1977 Jun;49(6):601-4. doi: 10.1093/bja/49.6.601. PMID 326281
- [Result] Friedman EA, Niswander KR, Sachtleben MR. Effect of diazepam on labor. Obstet Gynecol. 1969 Jul;34(1):82-6. No abstract available. PMID 4893003